CLINICAL TRIAL: NCT03893799
Title: A Phase 1b Dose-escalating Study With RBT-1 in Healthy Volunteers and Subjects With Stage 3/4 Chronic Kidney Disease
Brief Title: A Study of RBT-1 in Healthy Volunteers and Subjects With Stage 3/4 Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REN-001A
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 9 mg SnPP/240 mg FeS (Experimental)
  Interventions: Drug: RBT-1
- 27 mg SnPP/240 mg FeS (Experimental)
  Interventions: Drug: RBT-1
- 45 mg SnPP/240 mg FeS (Experimental)
  Interventions: Drug: RBT-1
- 63 mg SnPP/240 mg FeS (Experimental)
  Interventions: Drug: RBT-1
- 90 mg SnPP/240 mg FeS (Experimental)
  Interventions: Drug: RBT-1

INTERVENTIONS:
Drug: RBT-1 — Single intravenous administration

SUMMARY:
This is a Phase 1b, single-center, dose-escalating study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic effect of RBT-1 in healthy volunteers and in subjects with Stage 3/4 CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 80 years (inclusive, at time of ICF).
2. Body weight <125 kg.
3. Able and willing to comply with all study procedures.
4. Female subjects must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until 28 days after study drug administration.

   Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until 28 days after study drug administration. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
5. CKD Stage 3 as determined by estimated glomerular filtration rate (eGFR) between 30-59 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
6. CKD Stage 4 as determined by eGFR between 15-29 mL/min/1.73 m2 using the CKD-EPI equation.

Exclusion Criteria:

1. History of malignancy except carcinoma in situ in the cervix, early stage prostate cancer or non-melanoma skin cancers.
2. Use of investigational drugs or participation in another clinical trial within 30 days or 5 half-lives prior to screening, whichever is longer.
3. Serum ferritin > 500 ng/ml or who have received IV iron within 28 days of screening, or currently being treated with oral iron.
4. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
5. Any significant acute or chronic diseases.
6. Subjects with abnormal baseline liver tests or hepatitis serologies that suggest active infection.
7. Regular use of drugs of abuse and/or positive findings on urinary drug screening.
8. Current tobacco use and/or positive findings on urinary cotinine screening.
9. Subjects who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the subjects' tasks associated with the protocol.
10. Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
11. Subjects with history of photosensitivity or active skin disease
12. Known hypersensitivity or previous anaphylaxis to RBT-1 or to components thereof.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside Clinical Research, Edgewater, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zager RA, Johnson ACM, Guillem A, Keyser J, Singh B. A Pharmacologic "Stress Test" for Assessing Select Antioxidant Defenses in Patients with CKD. Clin J Am Soc Nephrol. 2020 May 7;15(5):633-642. doi: 10.2215/CJN.15951219. Epub 2020 Apr 14. PMID 32291269

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was pre-specified to analyze healthy volunteers and participants with CKD Stage 3/Stage 4 together and report results by dose.
Groups:
- 9 mg SnPP/240 mg FeS; 27 mg SnPP/240 mg FeS; 45 mg SnPP/240 mg FeS; 63 mg SnPP/240 mg FeS; 90 mg SnPP/240 mg FeS: Single IV infusion
Period: Overall Study
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS
Started | 6 | 18 | 6 | 6 | 18
Completed | 6 | 18 | 6 | 6 | 18
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS | Total
Number analyzed (Participants) | 6 | 18 | 6 | 6 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.75) | 60.0 (17.60) | 72.8 (4.54) | 71.8 (6.34) | 58.7 (20.08) | 61.0 (17.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 1 | 5 | 7 | 22
  Male | 6 | 9 | 5 | 1 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 6 | 15 | 6 | 6 | 17 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 1 | 6 | 14
  White | 3 | 11 | 6 | 5 | 11 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 1 | 4
Weight [Mean (Standard Deviation); unit: kg] | 93.3 (16.37) | 90.3 (16.8) | 92.9 (17.2) | 88.4 (17.18) | 82.9 (15.69) | 88.2 (16.34)
Height [Mean (Standard Deviation); unit: cm] | 180.9 (7.27) | 167.6 (9.26) | 166.4 (6.93) | 170.3 (7.41) | 168.5 (6.93) | 169.5 (8.66)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (4.61) | 32.3 (6.61) | 33.4 (4.77) | 30.7 (7.24) | 29.2 (5.63) | 30.8 (6.02)

OUTCOME MEASURES:

1. Primary Outcome: Effect of RBT-1 on Plasma Ferritin Levels
Time Frame: 24 hours post-infusion
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS
Number analyzed (Participants) | 6 | 18 | 6 | 6 | 18
Percent change from baseline | 592.3 [255.2 to 929.3] | 538.8 [345.1 to 732.5] | 313.7 [-23 to 650.4] | 308.2 [-27.6 to 644] | 610.9 [417.2 to 804.6]

2. Primary Outcome: Effect of RBT-1 on Plasma HO-1 Levels
Time Frame: 24 hours post-infusion
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS
Number analyzed (Participants) | 6 | 18 | 6 | 6 | 18
Percent change from baseline | -10.5 [-93.2 to 72.2] | 21 [-26.7 to 68.7] | 35.4 [-47.3 to 118] | 27.7 [-55.4 to 110.7] | 44.8 [-3.1 to 92.8]

3. Primary Outcome: Effect of RBT-1 on Plasma IL-10 Levels
Time Frame: 24 hours post-infusion
Population: Values at either baseline and/or the 24 h timepoint were missing from each of the treatment groups
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS
Number analyzed (Participants) | 1 | 4 | 6 | 2 | 6
Percent change from baseline | 66.8 [-715.9 to 849.5] | 95.5 [-323.5 to 514.5] | 574.6 [248.2 to 901.1] | 333.5 [-219.2 to 886.2] | 201.4 [-117.6 to 520.3]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | 9 mg SnPP/240 mg FeS | 27 mg SnPP/240 mg FeS | 45 mg SnPP/240 mg FeS | 63 mg SnPP/240 mg FeS | 90 mg SnPP/240 mg FeS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/18 | 0/6 | 0/6 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/18 | 0/6 | 0/6 | 0/18
Other Adverse Events (participants affected / at risk) | 0/6 | 6/18 | 1/6 | 5/6 | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9 mg SnPP/240 mg FeS (N=6) | 27 mg SnPP/240 mg FeS (N=18) | 45 mg SnPP/240 mg FeS (N=6) | 63 mg SnPP/240 mg FeS (N=6) | 90 mg SnPP/240 mg FeS (N=18)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Administration site discoloration (General disorders) | 0 | 0 | 0 | 0 | 2
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0
Infusion site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Injection site extravasation (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0
Hemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Bacteriuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 10
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03893799/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03893799/SAP_001.pdf